CLINICAL TRIAL: NCT06856967
Title: Evaluation of the Effect of Nirsevimab on Hospitalizations Due to RSV Infection in Infants Under One Year of Age: A Case-Control Study
Brief Title: Evaluation of the Effect of Nirsevimab on Hospitalizations Due to RSV Infection in Infants Under One Year of Age.
Status: Recruiting | Type: Observational
Sponsor: Meyer Children's Hospital IRCCS (Other)
Responsible Party: Principal Investigator, Giuseppe Indolfi, MD, Meyer Children's Hospital IRCCS
Other Study IDs: RAENHoB
Record Dates: First submitted 2025-02-26; First posted 2025-03-04 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2025-03

CONDITIONS: Respiratory Synctial Virus Infections
MeSH Terms: interventions — nirsevimab

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Cases: Patients aged <1 years hospitalized with confirmed bronchiolitis
  Interventions: Drug: Nirsevimab
- Controls: Patients aged <1 years hospitalized for condition other than confirmed bronchiolitis
  Interventions: Drug: Nirsevimab

INTERVENTIONS:
Drug: Nirsevimab — Evaluation of drug exposure in cases and controls

SUMMARY:
This study aims to evaluate the impact of Nirsevimab, a monoclonal antibody used for RSV prophylaxis, on reducing RSV- related hospitalizations. It will be conducted at 8 pediatric departments in Tuscany, Italy. First, a matched case-control study investigates the real-world effectiveness of Nirsevimab in preventing RSV-related lower respiratory tract infection (LRTI) hospitalizations during the RSV epidemic season 2024-2025. Second, a descriptive study examines how the Nirsevimab immunization campaign affects RSV epidemiology, focusing on patients' age, comorbidities, infection severity, and clinical outcomes. The findings aim to optimize RSV prevention strategies and inform public health policies.

ELIGIBILITY:
Inclusion Criteria:

Case patients

* Age <12 months
* Diagnosis of LRTI (i.e., bronchiolitis and/or pneumonia) at admission
* Positive RSV PCR on nasopharyngeal swab Control patients
* Age <12 months
* Diagnosis of LRTI (i.e., bronchiolitis and/or pneumonia) at admission
* Hospitalized for conditions other than respiratory infections

Exclusion Criteria:

* Parental refusal
* Previous immunization with Palivizumab
* Previous maternal RSV vaccine immunization during pregnancy

Max Age: 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Infants < 12 months during RSV 2024-2025 epidemic season
Sampling Method: Non-Probability Sample
Enrollment: 138 (Estimated)
Dates: Start 2024-12-04 (Actual); Primary Completion 2025-03 (Estimated); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
The proportion of patients immunized with Nirsevimab among children hospitalized for RSV-related LRTI and those in the control group. | November 2024-March 2025

CONTACTS AND LOCATIONS:
Locations (8):
- Italy (8):
  - SOC Pediatria Ospedale San Donato, Arezzo, Arezzo
  - SOC Pediatria Ospedale Santa Maria Annunziata, Bagno a Ripoli, Firenze
  - SOC Neonatologia e Terapia Intensiva Neonatale, Ospedale San Giovanni Di Dio, Florence, Firenze
  - Meyer Children's Hospital IRCCS, Florence, Italy
  - Azienda Ospedaliero Universitaria Pisana, Pisa, Italy
  - SOC Pediatria e Neonatologia Ospedale San Jacopo, Pistoia, Pistoia
  - SOC Pediatria e Neonatologia Ospedale Santo Stefano, Prato, Prato
  - SOC Pediatria AOU Senese, Siena, Siena